CLINICAL TRIAL: NCT04199546
Title: Chewing and Swallowing Training Program in Coffin-Lowry Syndrome: A Case Report
Brief Title: Chewing and Swallowing Training Program in Coffin-Lowry Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe Kübra Şahan, Principal investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA-94678
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Swallowing Disorder; Chewing Problem
MeSH Terms: conditions — Deglutition Disorders | interventions — Mastication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A child with Coffin-Lowry Syndrome (Other): A boy with a known CLS diagnosis with a history of coughing during eating, long-lasting wheezing, sputum and inability to intake solid food will be included.
  Interventions: Other: Chewing and swallowing rehabilitation

INTERVENTIONS:
Other: Chewing and swallowing rehabilitation — A home based chewing and swallowing training program (CST) will be applied by an experienced physical therapist. The Functional Chewing Training will be used to improve chewing function which has five steps including positioning the child and food, sensory stimulation, chewing training and adjustment of food consistency to improve chewing function. To support hyolaryngeal elevation, laryngeal mobilization will be performed. Hyolaryngeal mobilization will be performed by moving hyolaryngeal complex in right, left and up directions manually.

SUMMARY:
This study will report the chewing and swallowing disorders of a Coffin-Lowry Syndrome (CLS) patient, and effects of chewing and swallowing training on chewing and swallowing function.

DETAILED DESCRIPTION:
Patients with CLS suffer from spinal deformities, nonconvulsive status epilepticus, obstructive sleeep apnea syndrome, pneumonia, stimulus-induced myoclonus, cases of falls, mechanical ventilation, restrictive lung disease. It was also reported that patients with CLS had problems with eating and feeding functions. However there is no study investigating chewing and swallowing functions of this patient population. Therefore, the investigators have three main purposes:

1. To chewing and swallowing function in a boy with CLS diagnosis who was referred due to coughing during eating, long-lasting wheezing, sputum and inability to intake solid food
2. To investigate the effects of two months of chewing and swallowing training program
3. To present long term follow-up effects on chewing and swallowing function.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of CLS
* Having a history of coughing during eating, long-lasting wheezing, sputum
* Inability to intake solid food.

Exclusion Criteria:

- No history of coughing during eating, long-lasting wheezing, sputum

Ages: 3 Years to 3 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Instrumental swallowing evaluation | 6 months
  Videofluoroscopic Swallowing Evaluation (VFSE) will be performed. The swallowing physiology will be evaluated by using 3 ml of liquid and pudding barium during the VFSE. The Penetration and Aspiration Scale (PAS) will be used to determine penetration and aspiration severity, which is scored between 1 to 8. The score of PAS 1 means 'No aspiration', scores from 2 to 5 indicate 'Penetration', and scores from 6 to 8 indicate 'Aspiration'. High score indicates bad situation.

SECONDARY OUTCOMES:
Swallowing screening | 6 months
  The Pediatric Eating Assessment Tool (PEDI-EAT-10) instrument which has 10 questions to evaluate dysphagia symptom severity in children will be completed.
  Total scoring ranges from 0 to 40. Higher scores mean worse outcome.
Chewing evaluation | 6 months
  Karaduman Chewing Performance Scale will be used to define chewing performance level. It is a 5 point scale between 0 to 4. Level 0 means 'Normal chewing function', and level 4 means 'No biting and chewing'. Higher scores mean worse chewing function.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞE KÜBRA ŞAHAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)